CLINICAL TRIAL: NCT03635580
Title: Phase 2 Study of Efficacy and Safety of rhGH (Jintropin®) in Pediatric Participants With ISS (Idiopathic Short Stature): a 52-week Multicenter, Open-label, Randomized, Negative Controlled Study Followed by a 52-week Open-label Period
Brief Title: Efficacy and Safety of rhGH (Jintropin®) in Pediatric Participants With ISS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: The Children's Hospital of Zhejiang University School of Medicine (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Henan Provincial People's Hospital (Other); Children's Hospital of Fudan University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Shanxi Provincial Maternity and Children's Hospital (Other); The First Hospital of Jilin University (Other); Shanghai Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenSci 046 CT
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Dwarfism
MeSH Terms: conditions — Dwarfism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rhGH/Jintropin AQ (Experimental): Jintropin AQ, injection, 30IU/10mg/3ml/cartridge, 0.05mg /kg/d in phase 1 and 0.05-0.07mg/kg/d in phase 2.
  Interventions: Other: Negative control

INTERVENTIONS:
Other: Negative control — Untreated-control group

SUMMARY:
Phase 1: To evaluate the safety and efficacy of 0.05mg/kg/d of rhGH (Jintropin®) in the treatment of children with idiopathic short stature (ISS) in 52 weeks.

Phase 2: To evaluate the safety and efficacy of rhGH (Jintropin®) in the treatment of children with ISS in 2 years

ELIGIBILITY:
Inclusion Criteria:

* Boys are between 4 and 10 years old age and girls are between 4 and 9 years old age;
* Height <-2.25 SD (Standard deviation) for chronological age;
* GH (Growth hormone) peak concentration ≥10.0 ng/mL in GH stimulation tests;
* The bone age (BA) ≤chronological age (CA)+6 months;
* Prepubertal Status (Tanner Stage I);
* Birth weight within the normal range;
* Growth hormone treatment-naive;
* Participants are willing and able to cooperate to complete scheduled visits, treatment plans and laboratory tests and other procedures, to sign informed consent.

Exclusion Criteria:

* Participants with abnormal liver and kidney functions (ALT > upper limit 1.5 times of normal value; Cr > upper limit of normal value);
* Participants are positive for anti-HBc, HbsAg or HbeAg in Hepatitis B virus tests;
* Participants with known highly allergic constitution or allergy to investigational product or its excipient;
* Participants with systemic chronic disease and immune deficiency;
* Participants diagnosed with tumor, or with potential high tumor risks such as tumor markers exceed normal range and some other relative information may be excluded from the treatment;
* Participants with mental disease;
* Participants with other types of abnormal growth and development;

  1. Growth hormone deficiency (GHD) (confirmed by GH stimulation test);
  2. Turner syndrome (confirmed by karyotype test of girls);
  3. Noonan syndrome (hypertelorism, pectus carinatum, hypophrenia, frequently with skin disease and congenital heart disease, missense mutation of the protein tyrosine phosphatase, non-receptor type 11 (PTPN11) gene on chromosome 12 for half of the participants, for both male and female participants);
  4. Laron syndrome (confirmed by IGF-1 generation test);
  5. Small for gestational age ( the birth height or weight is below the tenth percentile or 2 SD, with catch-up growth uncompleted at 2 years old);
  6. Growth disorders caused by malnutrition or hypothyroidism (thyroid function test).
* Participants with impaired glucose regulation (IGR) (including impaired fasting glucose (IFG) and/or impaired glucose tolerance (IGT) ) or diabetes;
* BMI (Body mass index) ≥22kg/m²;
* Congenital skeletal abnormalities or scoliosis, claudication;
* Participants who took part in other clinical trials within 3 months;
* Participants who received medications which may interfere GH secretion or GH function, or other hormones within 3 months (such as sex steroids, glucocorticoids, etc.);
* Other conditions which is inappropriate for this study in the opinion of the investigator.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2018-06-11 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
ΔHtSDSca (The change of height standard deviation score of chronological age before and after treatment) | Baseline, 4,13,26,39,52,65,78,91,104 weeks after initiating treatment, 52 weeks in phase 1; 2 years in phase 2.
  ΔHtSDSca was the difference of HtSDSca before and after treatment, and HtSDSca was calculated by dividing the difference between the actual height of a patient and the mean height of the population for that chronological age by the standard deviation (SD) of the height of the population for that chronological age.

SECONDARY OUTCOMES:
ΔHT (Change of height) | Baseline, 4,13,26,39,52,65,78,91,104 weeks after initiating treatment, 52 weeks in phase 1; 2 years in phase 2.
△BA/CA (bone age change / chronological age) | Baseline, 4,13,26,39,52,65,78,91,104 weeks after initiating treatment, 52 weeks in phase 1; 2 years in phase 2.
Yearly growth velocity | Baseline, 4,13,26,39,52,65,78,91,104 weeks after initiating treatment, 52 weeks in phase 1; 2 years in phase 2.
ΔIGF-1 SDS (Change of insulin-like growth factor 1 standard deviation score) | Baseline, 4,13,26,39,52,65,78,91,104 weeks after initiating treatment, 52 weeks in phase 1; 2 years in phase 2.

CONTACTS AND LOCATIONS:
Overall Officials: Junfen Fu, Doctor, Principal Investigator — The Children's Hospital of Zhejiang University School of Medicine
Locations (9):
- China (9):
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Henan Children's Hospital, Zhengzhou, Henan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Children's Hospital of Shanxi, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - The Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Children's Hospital of Fudan University, Shanghai
  - Children's Hospital of Shanghai, Shanghai

REFERENCES:
- [Derived] Yuan J, Fu J, Wei H, Zhang G, Xiao Y, Du H, Gu W, Li Y, Chen L, Luo F, Zhong Y, Gong H. A Randomized Controlled Phase 3 Study on the Efficacy and Safety of Recombinant Human Growth Hormone in Children With Idiopathic Short Stature. Front Endocrinol (Lausanne). 2022 Apr 29;13:864908. doi: 10.3389/fendo.2022.864908. eCollection 2022. PMID 35573994